CLINICAL TRIAL: NCT04517825
Title: IGHID 11920 - More Than a Machine: Exploring the Ancillary Systems and Processes Required to Make Point-of-care HIV-1 Viral Load Testing Effective in Rural Western Uganda
Brief Title: More Than a Machine: Make Point-of-care HIV-1 Viral Load Testing Effective in Rural Uganda
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-2363; P30AI050410 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: HIV-1-infection
Keywords: viral load; CD4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Target Population: HIV positive individuals attending Bugoye ART clinic
  Interventions: Diagnostic Test: Cepheid Xpert HIV-1 Viral Load Assay

INTERVENTIONS:
Diagnostic Test: Cepheid Xpert HIV-1 Viral Load Assay — Rapid, on-site molecular HIV-1 viral load testing used in accordance with cleared/approved labeling

SUMMARY:
This is a two-phase study designed to assess measures of feasibility, sustainability, acceptability, penetration, and fidelity before and after implementation of a rapid molecular HIV-1 viral load testing infrastructure at a level III health center in rural western Uganda.

The central hypothesis is that implementation of PoC HIV-1 testing without accompanying modifications to clinic triage and flow, laboratory processes, and existing protocols guiding adherence counseling and regimen change, will not result in significant improvement in clinical outcomes in PLWH.

DETAILED DESCRIPTION:
This is a two-phase study designed to assess measures of feasibility, sustainability, acceptability, penetration, and fidelity before and after implementation of a rapid molecular HIV-1 viral load testing infrastructure at a level III health center in rural western Uganda.

In Phase 1, the study team will perform/record the following:

1. Administer a basic demographic and health questionnaire
2. Record routine clinical parameters during visit to include:

   1. Current ARV and prophylaxis regimen
   2. Last CD4 and VL, if available
   3. Clinical illness since last visit
3. Document the amount of time each patient spends in each phase of clinic (i.e. waiting room, provider, phlebotomy, waiting for results, adherence counseling).
4. Measure the number of participants requiring HIV-1 VL testing each clinic day, proportion electing to receive results by phone or at next visit.
5. Patients having blood drawn for HIV-1 VL testing will complete a semi-structured interview to explore perceptions of the current testing paradigm when results are received.
6. Provider and laboratory staff will complete a semi-structured interview to explore perceptions of the current testing paradigm with emphasis on workload

In Phase 2, the study team will perform/record the following:

1. Record routine clinical parameters during visit to include:

   1. Current ARV and prophylaxis regimen
   2. Last CD4 and VL, if available
   3. Clinical illness since last visit
2. Determine the amount of time each patient spends in each phase of clinic (i.e. waiting room, provider, phlebotomy, waiting for results, adherence counseling).
3. Measure the number of Xpert HIV-1 tests performed, the amount of time laboratory staff spends performing the tests and conducting maintenance, the number of tests failures and/or invalid tests, and equipment downtime related problems with software or power supply.
4. Measure the number of participants requiring HIV-1 VL testing each clinic day, proportion electing to receive results on same day, by phone, or next visit.
5. Patients having blood drawn for HIV-1 VL testing will complete a semi-structured interview to explore perceptions of the current testing paradigm when results are received.
6. Provider and laboratory staff will complete a semi-structured interview to explore perceptions of the current testing paradigm with emphasis on workload.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older receiving care at the Bugoye Health Center Antiretroviral therapy clinic

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years or older receiving care at the Bugoye Health Center Antiretroviral therapy clinic
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Tests Performed Successfully Each Clinic Day | Each clinic day for up to six months
  HIV viral load tests performed at peripheral health center
Number of Tests Performed Successfully each Month | Each month for up to six months
  HIV viral load tests performed at peripheral health center

SECONDARY OUTCOMES:
Proportion of Eligible Patients Electing to Stay to Receive Results | Each clinic day for up to six months
  Acceptability of rapid HIV viral load results
Proportion of Eligible Patients Electing to Stay to Receive Results | Each month for up to six months
  Acceptability of rapid HIV viral load results
Mean Time Clients Spend in Clinic | Each clinic day for up to 9 months
  Impact on routine ART Clinic flow
Provider Perception of Workload | Pre- and post-intervention (approximately 6 months apart)
  Perceived time spent conducting on-site testing vs send-out testing
Mean and median time-to-result | Up to 90 days after blood draw, after which considered not returned
  Mean and median number of days from blood draw to client receiving viral load result either from current standard of care or on-site testing
Machine Down-Time and Maintenance | Each clinic day (i.e. weekly) during the 6 months of Phase 2 when the Xpert is operational
  Total number of hours spent in maintenance, trouble-shooting, or repair

CONTACTS AND LOCATIONS:
Overall Officials: Ross M Boyce, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- Uganda (2):
  - Bugoye Level III Health Centre, Bugoye, Kasese
  - Mbarara University of Science and Technology (MUST), Mbarara

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: An investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Boyce RM, Ndizeye R, Ngelese H, Baguma E, Shem B, Rubinstein RJ, Rockwell E, Lotspeich SC, Shook-Sa BE, Ntaro M, Nyehangane D, Wohl DA, Siedner MJ, Mulogo EM. It takes more than a machine: A pilot feasibility study of point-of-care HIV-1 viral load testing at a lower-level health center in rural western Uganda. PLOS Glob Public Health. 2023 Mar 27;3(3):e0001678. doi: 10.1371/journal.pgph.0001678. eCollection 2023. PMID 36972208